CLINICAL TRIAL: NCT01497522
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study to Compare the Effect of 12 Weeks Treatment With LAF237 50 mg Bid to Placebo as Add-On Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Metformin Monotherapy
Brief Title: Efficacy and Safety of Vildagliptin as add-on Therapy to Metformin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLMF237A1301
Record Dates: First submitted 2011-12-20; First posted 2011-12-22 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Vildagliptin; Type 2 diabetes; HbA1c; Fasting plasma glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vildagliptin (Experimental): In addition to their stable dose of metformin monotherapy, patients should take vildagliptin 50 mg twice daily.
  Interventions: Drug: Vildagliptin
- Placebo (Placebo Comparator): In addition to their stable dose of metformin monotherapy, patients should take vildagliptin matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vildagliptin — vildagliptin 50 mg twice daily
  Other Names: LAF237
  Arms: Vildagliptin
Drug: Placebo — Matching Placebo of vildagliptin 50 mg twice daily
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of vildagliptin 50 mg bid as an add-on therapy to metformin in Japanese patients with T2DM. This study is being conducted to support registration of the fixed-dose combination of vildagliptin and metformin for the treatment of Type 2 diabetes mellitus (T2DM) in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes inadequately controlled with diet, exercise and oral anti-diabetic therapy.
* HbA1c in the range of 7.0-10.0%
* Body mass index in the range 20-35 kg/m2

Exclusion Criteria:

* Type 1 diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes
* Significant heart diseases

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin (HbA1c) at 12 weeks between treatment groups | Baseline to 12 weeks
  HbA1c will be performed on a blood sample obtained by study personnel and measured by high-performance liquid chromatography (HPLC) performed at a central laboratory.

SECONDARY OUTCOMES:
Change from baseline in HbA1c at 12 weeks within subgroups of metformin doses | Baseline to 12 weeks
  HbA1c will be performed on a blood sample obtained by study personnel and measured by high-performance liquid chromatography (HPLC) performed at a central laboratory.
Change from baseline in Fasting plasma glucose (FPG) at 12 weeks | Baseline to 12 weeks
  FPG will be performed on a blood sample obtained by study personnel and analyzed at a central laboratory.
Percentage of patients meeting Responder rates in HbA1c | 12 weeks
  Responder rates will be categorized by predefined HbA1c value at 12 weeks :
  * Endpoint HbA1c ≤ 6.5%
  * Endpoint HbA1c ≤ 7%
  * Endpoint HbA1c ≤ 7% in patients with baseline HbA1c ≤ 8%
Number of patients with adverse events (including hypoglycemia), serious adverse events and death | 12 weeks
  The occurrence of adverse events will be sought by non-directive questioning of the patient at each visit. Adverse events are defined as appearance or worsening of any undesirable symptom, sign (including an abnormal laboratory finding), or medical conditions. Serious adverse events are any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalization, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgment of investigators represent significant hazards.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- Japan (17):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kitakyushu, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Ohkawa-city, Fukuoka
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Takatsuki, Osaka
  - Novartis Investigative Site, Ageo, Saitama
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Edogawa-ku, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Kiyose, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Nerima-ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo

REFERENCES:
- [Result] Odawara M, Hamada I, Suzuki M. Efficacy and Safety of Vildagliptin as Add-on to Metformin in Japanese Patients with Type 2 Diabetes Mellitus. Diabetes Ther. 2014 Jun;5(1):169-81. doi: 10.1007/s13300-014-0059-x. Epub 2014 Mar 7. PMID 24604395